CLINICAL TRIAL: NCT07053150
Title: A Prospective, Open-label, Exploratory Basket Trial to Evaluate the Efficacy and Safety of Sintilimab Combined With Pyrotinib ± Chemotherapy in Patients With Advanced Digestive System Tumors (CCGLC-018)
Brief Title: A Prospective, Open-label, Exploratory Basket Trial to Evaluate the Efficacy and Safety of Sintilimab Combined With Pyrotinib ± Chemotherapy in Patients With Advanced Digestive System Tumors
Acronym: CCGLC-018
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Ze-yang Ding, MD, Prof., Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-S045
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Digestive System Tumor
Keywords: Pyrotinib; Sintilimab; HER2-Positive Advanced digestive system tumors; HER2-positive tumors; Immunotherapy; Targeted therapy
MeSH Terms: interventions — sintilimab; spartalizumab; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HER2-Positive Gastric Cancer (Experimental): Patients with HER2-positive advanced or metastatic gastric cancer will receive sintilimab (200 mg IV, Q3W) and pyrotinib (400 mg PO, QD), with or without chemotherapy. The investigator may choose from XELOX, SOX, or TS regimens based on clinical evaluation.
  Interventions: Drug: Sintilimab; Drug: Pyrotinib; Drug: Optional Chemotherapy
- HER2-Positive Colorectal Cancer (Experimental): Patients with HER2-positive advanced or metastatic colorectal cancer will receive sintilimab (200 mg IV, Q3W) and pyrotinib (400 mg PO, QD), with or without chemotherapy. The recommended regimens include mFOLFOX6 or XELOX, at the investigator's discretion.
  Interventions: Drug: Sintilimab; Drug: Pyrotinib; Drug: Optional Chemotherapy
- HER2-Positive Hepatocellular Carcinoma (Experimental): Patients with HER2-positive advanced or unresectable hepatocellular carcinoma will receive sintilimab (200 mg IV, Q3W) and pyrotinib (400 mg PO, QD), with or without chemotherapy. Chemotherapy may include FOLFOX or interventional locoregional therapies, as appropriate.
  Interventions: Drug: Sintilimab; Drug: Pyrotinib; Drug: Optional Chemotherapy
- HER2-Positive Biliary Tract Cancer (Experimental): Patients with HER2-positive advanced or metastatic biliary tract cancer (including intrahepatic and extrahepatic cholangiocarcinoma, gallbladder cancer) will receive sintilimab (200 mg IV, Q3W) and pyrotinib (400 mg PO, QD), with or without chemotherapy. Suggested regimens include GC (gemcitabine + cisplatin) or GEMOX.
  Interventions: Drug: Sintilimab; Drug: Pyrotinib; Drug: Optional Chemotherapy
- HER2-Positive Pancreatic Cancer (Experimental): Patients with HER2-positive advanced or metastatic pancreatic cancer will receive sintilimab (200 mg IV, Q3W) and pyrotinib (400 mg PO, QD), with or without chemotherapy. Optional chemotherapy regimens include FOLFIRINOX or AG (nab-paclitaxel + gemcitabine).
  Interventions: Drug: Sintilimab; Drug: Pyrotinib; Drug: Optional Chemotherapy

INTERVENTIONS:
Drug: Sintilimab — Dosage Form: Intravenous (IV) infusion Dosage: 200 mg Frequency: Every 3 weeks (Q3W) Duration: Until disease progression, unacceptable toxicity, or up to 2 years
  Other Names: Anti-PD-1 Monoclonal Antibody
Drug: Pyrotinib — Dosage Form: Oral tablet Dosage: 400 mg once daily (QD) Frequency: Continuous daily dosing Duration: Until disease progression or intolerable toxicity
  Other Names: Pan-HER Tyrosine Kinase Inhibitor
Drug: Optional Chemotherapy — 1. FOLFOX:
     Oxaliplatin 85 mg/m² IV Day 1, leucovorin 400 mg/m² IV Day 1, 5-FU 400 mg/m² IV bolus + 2400 mg/m² continuous infusion over 46h (Days 2-3)
  2. GEMOX:
     Gemcitabine 1000 mg/m² and oxaliplatin 100 mg/m² IV Day 1
  3. GC:
     Gemcitabine 1000 mg/m² and cisplatin 25 mg/m² IV on Days 1 and 8
  4. XELOX (CapeOX) Oxaliplatin 130 mg/m² IV Day 1, capecitabine 1000 mg/m² PO BID Days 1-14
  5. SOX:
     Oxaliplatin 130 mg/m² IV Day 1, S-1 PO BID Days 1-14 (dose based on BSA: <1.25 m² = 40 mg, 1.25-<1.5 m² = 50 mg, ≥1.5 m² = 60 mg)
  6. TS:
     Paclitaxel 80 mg/m² IV Days 1 and 8, S-1 as above
  7. mFOLFOX6: Same as FOLFOX; used primarily in colorectal cancer
  8. FOLFIRINOX:
     Leucovorin 400 mg/m², 5-FU (bolus + continuous), irinotecan 180 mg/m², oxaliplatin 85 mg/m² IV Day 1
  9. AG:
  Nab-paclitaxel 125 mg/m² and gemcitabine 1000 mg/m² IV on Days 1 and 8

SUMMARY:
This is a prospective, open-label, exploratory, phase II basket clinical trial designed to evaluate the efficacy and safety of sintilimab in combination with pyrotinib with or without chemotherapy in patients with advanced HER2-positive digestive system malignancies. Eligible patients include those with locally advanced unresectable or metastatic gastric, colorectal, hepatocellular, biliary tract, or pancreatic cancers. Patients will receive sintilimab and pyrotinib, with chemotherapy regimens selected at the investigator's discretion based on tumor type and clinical condition. The primary endpoint is objective response rate (ORR), with secondary endpoints including progression-free survival (PFS), disease control rate (DCR), overall survival (OS), and safety.

DETAILED DESCRIPTION:
Immunotherapy, particularly immune checkpoint inhibitors (ICIs), has significantly advanced the treatment landscape for various solid tumors, but many patients still fail to respond or develop resistance. Combining ICIs with targeted agents may overcome these limitations. Pyrotinib is a pan-ErbB irreversible tyrosine kinase inhibitor (TKI) with potent activity against HER2, which is overexpressed in multiple digestive tract cancers including gastric, colorectal, biliary tract, and pancreatic cancers.

This basket trial investigates the efficacy and safety of sintilimab (a PD-1 inhibitor) combined with pyrotinib, with or without chemotherapy, in HER2-positive digestive system tumors. Patients must meet HER2 positivity criteria via IHC, FISH/CISH, or NGS. The study uses a Bayesian adaptive design to independently evaluate efficacy across cancer subtypes.

Patients will receive sintilimab (200 mg IV every 3 weeks) and pyrotinib (400 mg orally daily). Chemotherapy is optional and tailored by tumor type, including regimens such as FOLFOX, GC, XELOX, or AG, among others.

Primary endpoint: ORR per RECIST 1.1. Secondary endpoints: PFS, DCR, OS, and treatment-related adverse events (TRAEs).

The total planned enrollment is approximately 80 patients, with flexible sample size adjustments based on interim Bayesian analysis within each tumor cohort. Exploratory objectives include biomarker analysis (e.g., PD-L1, TMB, HER2 amplification/mutation) and tumor microenvironment changes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with unresectable locally advanced T3-4 stage or M1 stage metastatic digestive system tumors confirmed by histology or cytology, including gastric cancer, colorectal cancer, hepatocellular carcinoma, biliary tract cancer and pancreatic cancer
* Patients who have not received systematic treatment in the past or whose disease has progressed or is intolerant after standard first-line treatment, and whose disease has progressed for more than 6 months after neoadjuvant therapy/whose last adjuvant therapy failed/who have completed (new) adjuvant therapy for less than 6 months from disease recurrence can be enrolled
* Histologically or cytologically confirmed HER2-positive (IHC 3+ or IHC 2+/FISH-amplified/NGS-confirmed) locally advanced or metastatic digestive system tumors (including gastric, colorectal, hepatocellular, biliary tract cancers)
* ECOG performance status 0-2
* At least one measurable lesion per RECIST 1.1 criteria
* Adequate organ function:
* Hematologic: ANC ≥1.5×10⁹/L, platelets ≥75×10⁹/L, hemoglobin ≥9 g/dL
* Hepatic: Total bilirubin ≤1.5×ULN; ALT/AST ≤2.5×ULN (≤5×ULN for liver metastases/HCC); albumin ≥28 g/L
* Renal: Serum creatinine ≤1.5×ULN or CrCl ≥50 mL/min; urine protein <2+ (if ≥2+, 24-hour urine protein <1 g)
* Coagulation: INR ≤2.3 or PT prolongation ≤6 seconds
* Life expectancy ≥12 weeks
* Fertile patients must use effective contraception during treatment and for 6 months after last dose
* Willing and able to provide written informed consent

Exclusion Criteria:

* Previous treatment with any HER2-targeted therapy (e.g., trastuzumab)
* History of hematologic malignancies
* Pregnancy, lactation, or plans to become pregnant during study
* Last anticancer therapy ≤28 days prior to enrollment or unresolved toxicities from prior therapy
* Contraindications to immunotherapy including:
* History of organ transplantation
* Severe autoimmune diseases
* Grade ≥4 immune-related adverse events from prior immunotherapy
* Uncontrolled active infections
* Use of systemic immunosuppressants (>10 mg/day prednisone equivalent) within 14 days
* Known hypersensitivity to PD-1 inhibitors, pyrotinib, or monoclonal antibodies
* Participation in other clinical trials within 3 months
* Symptomatic ascites, pleural or pericardial effusion requiring drainage
* Life-threatening bleeding events within 3 months or arterial/venous thrombosis within 6 months (except stable catheter-related thrombosis)
* History of pulmonary fibrosis, interstitial lung disease, or drug-related pneumonitis
* Active tuberculosis requiring treatment or treated within past year
* Major surgery within 4 weeks or unhealed surgical wounds
* Severe dysfunction of major organs (heart, lungs, liver, kidneys, CNS)
* Any other condition that may increase risk or interfere with study results as judged by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months.
  Proportion of patients achieving complete response (CR) or partial response (PR) as assessed by investigators according to RECIST v1.1. Responses must be confirmed by repeat imaging ≥4 weeks (±7 days) after the initial documentation.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 36 months.
  Time from initiation of treatment to the first documentation of disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 24 months.
  Proportion of patients who achieve CR, PR, or stable disease (SD) as the best overall response per RECIST v1.1.
Overall Survival (OS) | Up to 36 months.
  Time from treatment initiation to death from any cause. Patients who are alive at the last follow-up will be censored at the date of last contact.
Treatment-Related Adverse Events (TRAEs) | From first dose through 90 days after last dose.
  Incidence, severity, and type of treatment-related adverse events as assessed by NCI-CTCAE v5.0, including laboratory abnormalities and dose interruptions or discontinuations due to toxicity.

OTHER OUTCOMES:
Biomarker Analysis (PD-L1, TMB, HER2 Amplification) | Baseline (pre-treatment) and at time of disease progression (if re-biopsied), assessed up to 36 months.
  Correlation between biomarker status (e.g., PD-L1 expression, tumor mutational burden) and treatment response.
Tumor Microenvironment Changes (CD8+ T Cells, Tregs) | Baseline (pre-treatment) and at time of disease progression (if re-biopsied), assessed up to 36 months.
  Immunohistochemical analysis of pre- and post-treatment tumor immune infiltrates.

CONTACTS AND LOCATIONS:
Overall Officials: Ze-yang Ding, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China